CLINICAL TRIAL: NCT00357071
Title: Evaluation of Immune Responses to Different Antigens in Non Infectious Ocular Inflammatory Diseases
Brief Title: Immune Responses to Antigens in Non-infectious Eye Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030122; 03-EI-0122
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07-24

CONDITIONS: Eye Diseases
Keywords: Autoimmunity; Cell Mediated Immunity; S Antigen; Cell Proliferation; Uveitis; Cell Proliferation Assays; Auto-Antibody; Auto-Antigens
MeSH Terms: conditions — Eye Diseases; Autoimmune Diseases; Hyperplasia; Uveitis

SUMMARY:
This study will collect blood samples from patients with non-infectious eye inflammatory diseases a spectrum of eye disorders that can produce sight-threatening vision loss. The blood will be analyzed for substances that may provide a better understanding of the nature of these disorders, possibly leading to improved treatments. Treatment is not offered under this protocol.

Patients 6 years of age and older with an eye inflammatory disease, including non-infectious uveitis, ocular cicatricial pemphigoid, non-infectious scleritis, episcleritis, Stevens Johnson syndrome, Moorens ulcer, peripheral ulcerative keratitis and keratoconjunctivitis sicca, may be eligible for this study. Patients may or may not currently be participating in a treatment trial.

Participants will have blood drawn through a needle in an arm vein. More samples may be collected if patients enrolled in another study are scheduled for additional visits. No more than 4 teaspoonfuls of blood will be collected at any one time.

DETAILED DESCRIPTION:
Ocular inflammatory diseases can lead to visual loss in adults as well as in children. These conditions are usually characterized by repeated exacerbations and remissions. The underlying cause of majority of these conditions is not clear even though an autoimmune mechanism has been implicated. Various studies have reported an altered immunological profile in these patients. An underlying immune mechanism has been thought to be playing a role in at least some of the ocular inflammatory diseases. In addition, evidence from literature also suggests inflammatory disease may be an important mechanism leading to Age related macular degeneration and Diabetic retinopathy, two leading causes for vision loss. However, very little is known about the involvement of immune components in these patients.

This protocol proposes to test for proliferative cell mediated and humoral responses against self-antigens from patients with ocular inflammatory diseases, AMD and diabetic retinopathy. Patients will be recruited from other ongoing protocols. An attempt would be made to find any correlation between the clinical disease and the immunological findings. These findings will not be used for diagnostic nor therapeutic purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant is 6 years or older.
  2. Adult participant is able to understand and sign the informed consent. If the participant is younger than 18 years of age at enrollment, has a parent or legal guardian who is able to understand and sign the consent on their behalf. Children must provide assent.
  3. Patients must have a diagnosis of an ocular inflammatory disease, AMD or diabetic retinopathy.

EXCLUSION CRITERIA:

1. The presence of non-ocular inflammatory disease.
2. Unwilling or unable to provide a blood sample.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2003-04-07; Study Completion 2018-07-24

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Foster CS, Kenyon KR, Greiner J, Greineder DK, Friedland B, Allansmith MR. The immunopathology of Mooren's ulcer. Am J Ophthalmol. 1979 Aug;88(2):149-59. doi: 10.1016/0002-9394(79)90459-8. PMID 382859
- [Background] Kriukova ME, Bocharova-Messner OM, Stefanov SB. [Shape factor of myofibril cross sections of functionally different muscles of the cricket Acheta domestica]. Zh Evol Biokhim Fiziol. 1978 Nov-Dec;14(6):571-5. No abstract available. Russian. PMID 735597
- [Background] Murray PI, Rahi AH. Pathogenesis of Mooren's ulcer: some new concepts. Br J Ophthalmol. 1984 Mar;68(3):182-7. doi: 10.1136/bjo.68.3.182. PMID 6230102